CLINICAL TRIAL: NCT02141516
Title: A Phase IIIb, Open Label, Controlled, Multi-Center Study to Evaluate the Safety, Tolerability and Immunogenicity of Two Doses of Novartis Meningococcal Group B Vaccine When Administered to Immunocompromised Patients From 2 to 17 Years of Age Who Are at Increased Risk of Meningococcal Disease Because of Complement Deficiency or Asplenia Compared to Matched Healthy Controls.
Brief Title: Safety and Immunogenicity of Novartis Meningococcal B Vaccine When Administered to Immunocompromised Children and Adolescents Compared to Healthy Subjects.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V72_62; 2013-002454-78 (EudraCT Number)
Record Dates: First submitted 2014-05-15; First posted 2014-05-19 (Estimated); Results first posted 2017-02-15 (Actual); Last update posted 2017-02-15 (Actual); Status verified 2016-07

CONDITIONS: Meningococcal Disease
Keywords: Meningitis; vaccination; complement deficiency; asplenia; splenic dysfunction
MeSH Terms: conditions — Meningococcal Infections; Meningitis; Hereditary Complement Deficiency Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A (Experimental): Complement deficiency
  Interventions: Biological: rMenB+OMV
- Group B (Experimental): asplenia/splenic dysfunction
  Interventions: Biological: rMenB+OMV
- Group C (Active Comparator): age-matched healthy controls
  Interventions: Biological: rMenB+OMV

INTERVENTIONS:
Biological: rMenB+OMV — 2 doses of vaccine 2 months apart
  Arms: Group A
Biological: rMenB+OMV — 2 doses of vaccine 2 months apart
  Arms: Group B
Biological: rMenB+OMV — 2 doses of vaccine 2 months apart
  Arms: Group C

SUMMARY:
The study aims at evaluating the safety and immunogenicity of rMenB+OMV NZ when administered to subjects from 2 to 17 years of age with increased risk of meningococcal disease because either of primary or secondary complement deficiencies or of asplenia or splenic dysfunction. A group of healthy age-matched subjects will be enrolled to serve as a descriptive control for immunogenicity and safety.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criterion applicable to All Groups

* Subjects aged 2 to 17 years (inclusive) at enrollment
* weighing at least 13 Kg at the time of enrollment

Inclusion criterion applicable to Group A - Subjects at risk of meningococcal disease because of primary or secondary complement deficiencies

Inclusion criterion applicable to Group B

- Subjects at risk of meningococcal disease because of functional or anatomic asplenia

Inclusion criterion applicable to Group C - healthy subjects

Exclusion Criteria:

Exclusion criteria applicable to All Groups (A, B and C)

* History of any previous immunization with a meningococcal B vaccine
* History of severe allergic reaction after previous vaccinations, or hypersensitivity to any component of the vaccine
* Known HIV infection
* History of any progressive or severe neurologic disorder or seizure disorder
* Contraindication to intramuscular injection or blood drawn
* Females who are pregnant, planning a pregnancy or nursing (breastfeeding)
* Females of childbearing potential who have not used or do not plan to use acceptable birth control measures
* History or any illness/condition that, in the opinion of the investigator, might interfere with the results of the study or pose additional risk to the subjects

Exclusion criterion applicable to Groups A and B

- Previous known or suspected disease caused by N. meningitidis in the last year.

Exclusion criteria applicable to Group C

* Previous known or suspected disease caused by N. meningitidis
* Known or suspected impairment/alteration of the immune system

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 239 (Actual)
Dates: Start 2014-05; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis Vaccines
Locations (20):
- Italy (5):
  - 12, Novartis Investigational Site, Florence
  - 11, Novartis Investigational Site, Genova
  - 10, Novartis Investigational Site, Milan
  - 14, Novartis Investigational Site, Padua
  - 13, Novartis Investigational Site, Roma
- Poland (3):
  - 31, Novartis Investigational Site, Krakow
  - 33, Novartis Investigational Site, Warsaw
  - 30, Novartis Investigational Site, Wroclaw
- Russia (3):
  - 42, Novartis Investigational Site, Moscow
  - 41, Novartis Investigational Site, Moscow
  - 43, Novartis Investigational Site, Yekaterinburg
- Spain (5):
  - 21, Novartis Investigational Site, Barcelona
  - 22, Novartis Investigational Site, Madrid
  - 23, Novartis Investigational Site, Madrid
  - 20, Novartis Investigational Site, Santiago de Compostela
  - 24, Novartis Investigational Site, Valencia
- United Kingdom (4):
  - 53, Novartis Investigational Site, London
  - 52, Novartis Investigational Site, Manchester
  - 50, Novartis Investigational Site, Oxford
  - 51, Novartis Investigational Site, Southampton

REFERENCES:
- [Derived] Martinon-Torres F, Bernatowska E, Shcherbina A, Esposito S, Szenborn L, Marti MC, Hughes S, Faust SN, Gonzalez-Granado LI, Yu LM, D'Agostino D, Calabresi M, Toneatto D, Snape MD. Meningococcal B Vaccine Immunogenicity in Children With Defects in Complement and Splenic Function. Pediatrics. 2018 Sep;142(3):e20174250. doi: 10.1542/peds.2017-4250. Epub 2018 Aug 1. PMID 30068713

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at 4 centers in Italy, 3 centers in Poland, 3 centers in the Russian Federation, 4 centers in Spain and 4 centers in the United Kingdom.
Pre-assignment Details: All the enrolled subjects were included in the trial. One subject did not complete the study because he/she did not meet criteria for re-vaccination; two subjects met enrollment delay criteria since they required regular blood transfusions and they were unable to commit to visit windows (screen failure).
Groups:
- CompDef: Subjects aged ≥ 2 to ≤ 17 years with complement deficiencies received 2 doses of rMenB+OMV NZ administered 2 months apart.
- Asplenia: Subjects aged ≥ 2 to ≤ 17 years with Asplenia received 2 doses of rMenB+OMV NZ administered 2 months apart.
- Healthy: Healthy subjects aged ≥ 2 to ≤ 17 years received 2 doses of rMenB+OMV NZ administered 2 months apart.
Period: Overall Study
Arm/Group | CompDef | Asplenia | Healthy
Started | 40 | 112 | 87
Completed | 40 | 107 | 87
Not Completed | 0 | 5 | 0
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Other | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Asplenia: Subjects aged ≥ 2 to ≤17 years with Asplenia received 2 doses of rMenB+OMV NZ administered 2 months apart.
- Total: Total of all reporting groups
Arm/Group | CompDef | Asplenia | Healthy | Total
Number analyzed (Participants) | 40 | 112 | 87 | 239
Age, Continuous [Mean (Standard Deviation); unit: Years] | 8.5 (4.35) | 11.1 (3.7) | 10.2 (4.14) | 10.3 (4.07)
Sex/Gender, Customized [Number; unit: participants]
  Female | 17 | 46 | 44 | 107
  Male | 23 | 66 | 43 | 132

OUTCOME MEASURES:

1. Primary Outcome: Percentages of Subjects With Serum Bactericidal Activity Using Human Complement (hSBA) Titers ≥ 5 for B Indicator Strains (H44/76, 5/99, and NZ98/254) and M10713 Strain.
Description: Immunogenicity was assessed in terms of percentage of subjects with hSBA titers ≥ 5 against N. meningitidis serogroup B indicator strains (H44/76, 5/99, and NZ98/254) and M10713 strain following 2 doses of rMenB+Outer Membrane Vesicle (OMV) NZ, administered on Day 1 and Day 61.
Time Frame: Day 1 and Day 91 (one month after the second dose of the study vaccine)
Population: Analysis was done on Full Analysis Set (all subjects in the enrolled set who: received a study vaccination and provided an evaluable serum sample at 1 month after the second dose of rMenB+OMV NZ, with assay result available for at least one of the serogroup B indicator strains or M10713 strain or ELISA).
Measure: Number (95% Confidence Interval); unit: Percentage of Subjects
Groups:
- CompDef + Asplenia: Subjects aged ≥ 2 to ≤ 17 years with either complement deficiencies or Asplenia received 2 doses of rMenB+OMV NZ administered 2 months apart.
Arm/Group | CompDef | Asplenia | CompDef + Asplenia | Healthy
Number analyzed (Participants) | 39 | 106 | 145 | 85
Percentage of Subjects
  5/99 - Day 1 (N=37,103,140,82) | 0 [0 to 9.5] | 12 [6.2 to 19.5] | 9 [4.5 to 14.5] | 6 [2 to 13.7]
  5/99 - Day 91 (N=38,106,144,83) | 95 [82.3 to 99.4] | 100 [96.6 to 100] | 99 [95.1 to 99.83] | 99 [93.5 to 99.97]
  H44/76 - Day 1 (N=39,104,143,84) | 0 [0 to 9] | 7 [2.7 to 13.4] | 5 [2 to 9.8] | 6 [2 to 13.3]
  H44/76 - Day 91 (N=39,104,143,85) | 87 [72.6 to 95.7] | 97 [91.8 to 99.4] | 94 [89.3 to 97.6] | 98 [91.8 to 99.71]
  M10713 - Day 1 (N=36,102,138,82) | 56 [38.1 to 72.1] | 79 [70.3 to 86.8] | 73 [65 to 80.4] | 78 [67.5 to 86.4]
  M10713 - Day 91 (N=37,103,140,83) | 73 [55.9 to 86.2] | 94 [87.8 to 97.8] | 89 [82.1 to 93.3] | 99 [93.5 to 99.97]
  NZ98/254 - Day 1 (N=36,105,141,83) | 0 [0 to 9.7] | 4 [1 to 9.5] | 3 [0.8 to 7.1] | 2 [0.29 to 8.4]
  NZ98/254 - Day 91 (N=38,106,144,84) | 68 [51.3 to 82.5] | 86 [77.7 to 91.9] | 81 [73.9 to 87.3] | 83 [73.6 to 90.6]

2. Primary Outcome: Percentages of Subjects With hSBA Titers ≥ 8 for B Indicator Strains (H44/76, 5/99, and NZ98/254) and M10713 Strain.
Description: Immunogenicity was assessed in terms of percentage of subjects with hSBA titers ≥ 8 against N. meningitidis serogroup B indicator strains (H44/76, 5/99, and NZ98/254) and M10713 strain following 2 doses of rMenB+OMV NZ, administered on Day 1 and Day 61.
Time Frame: Day 1 and Day 91 (one month after the second dose of the study vaccine).
Population: Analysis was done on Full Analysis Set
Measure: Number (95% Confidence Interval); unit: Percentage of Subjects
Arm/Group | CompDef | Asplenia | CompDef + Asplenia | Healthy
Number analyzed (Participants) | 40 | 107 | 147 | 87
Percentage of Subjects
  5/99 - Day 1 (N=37,103,140,82) | 0 [0 to 9.5] | 11 [5.5 to 18.3] | 8 [4 to 13.6] | 5 [1.3 to 12]
  5/99 - Day 91 (N=38,106,144,83) | 92 [78.6 to 98.3] | 100 [96.6 to 100] | 98 [94 to 99.57] | 99 [93.5 to 99.97]
  H44/76 - Day 1 (N=39,104,143,84) | 0 [0 to 9] | 2 [0.23 to 6.8] | 1 [0.17 to 5] | 2 [0.29 to 8.3]
  H44/76 - Day 91 (N=39,104,143,85) | 87 [72.6 to 95.7] | 95 [89.1 to 98.4] | 93 [87.5 to 96.6] | 98 [91.8 to 99.71]
  M10713 - Day 1 (N=36,102,138,82) | 47 [30.4 to 64.5] | 68 [57.7 to 76.6] | 62 [53.7 to 70.4] | 68 [57.1 to 78.1]
  M10713 - Day 91 (N=37,103,140,83) | 70 [53 to 84.1] | 94 [87.8 to 97.8] | 88 [81.3 to 92.8] | 98 [91.6 to 99.71]
  NZ98/254 - Day 1 (N=36,105,141,83) | 0 [0 to 9.7] | 4 [1 to 9.5] | 3 [0.8 to 7.1] | 0 [0 to 4.3]
  NZ98/254 - Day 91 (N=38,106,144,84) | 63 [46 to 78.2] | 79 [70.3 to 86.5] | 75 [67.1 to 81.8] | 73 [61.8 to 81.8]

3. Primary Outcome: Geometric Mean Ratios (GMRs) Against N. Meningitidis Serogroup B Strains Following a 2-dose Vaccination Schedule.
Description: Immunogenicity was assessed in terms of GMRs against N. meningitidis serogroup B indicator strains (H44/76, 5/99, and NZ98/254) and M10713 strain following 2 doses of rMenB+OMV NZ, administered on Day 1 and Day 61.
Time Frame: Day 1 and Day 91 (one month after the second dose of the study vaccine).
Population: Analysis was done on Full Analysis Set
Measure: Geometric Mean (95% Confidence Interval); unit: Ratios
Arm/Group | CompDef | Asplenia | CompDef + Asplenia | Healthy
Number analyzed (Participants) | 40 | 107 | 147 | 85
Ratios
  5/99 - Day 91/Day 1 (N=37,103,140,82) | 299 [170 to 525] | 207 [149 to 288] | 228 [173 to 302] | 245 [187 to 321]
  H44/76 - Day 91/Day 1 (N=39,104,143,84) | 44 [27 to 73] | 56 [41 to 75] | 52 [41 to 67] | 66 [52 to 83]
  M10713 - Day 91/Day 1 (N=36,102,138,82) | 2.25 [1.37 to 3.71] | 2.95 [2.21 to 3.95] | 2.75 [2.15 to 3.51] | 2.71 [2.02 to 3.65]
  NZ98/254 - Day 91/Day 1 (N=36,105,141,83) | 8.58 [4.9 to 15] | 16 [12 to 22] | 14 [10 to 18] | 13 [10 to 17]

4. Primary Outcome: Geometric Mean hSBA Titers (GMTs) Against N. Meningitidis Serogroup B Strains Following a 2-dose Vaccination Schedule.
Description: Immunogenicity was assessed in terms of GMTs against N. meningitidis serogroup B indicator strains (H44/76, 5/99, and NZ98/254) and M10713 strain following 2 doses of rMenB+OMV NZ, administered on Day 1 and Day 61.
Time Frame: Day 1 and Day 91 (one month after the second dose of the study vaccine).
Population: Analysis was done on Full Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | CompDef | Asplenia | CompDef + Asplenia | Healthy
Number analyzed (Participants) | 40 | 107 | 147 | 85
Titers
  5/99 - Day 1 (N=37,103,140,82) | 0.87 [0.61 to 1.26] | 1.43 [1.16 to 1.78] | 1.26 [1.05 to 1.51] | 1.24 [1.02 to 1.52]
  5/99 - Day 91 (N=38,106,144,83) | 263 [166 to 415] | 300 [230 to 392] | 290 [231 to 362] | 307 [250 to 376]
  H44/76 - Day 1 (N=39,104,143,84) | 1.08 [0.87 to 1.33] | 1.17 [1.03 to 1.32] | 1.14 [1.03 to 1.26] | 1.15 [1.03 to 1.28]
  H44/76 - Day 91 (N=39,104,143,85) | 48 [29 to 79] | 65 [48 to 88] | 60 [46 to 77] | 76 [61 to 94]
  M10713 - Day 1 (N=36,102,138,82) | 8.57 [4.43 to 17] | 15 [10 to 22] | 13 [9.44 to 18] | 16 [11 to 22]
  M10713 - Day 91 (N=37,103,140,83) | 20 [11 to 34] | 45 [33 to 62] | 36 [28 to 47] | 42 [34 to 52]
  NZ98/254 - Day 1 (N=36,105,141,83) | 0.95 [0.78 to 1.16] | 1.1 [0.98 to 1.24] | 1.06 [0.96 to 1.17] | 1.05 [0.98 to 1.12]
  NZ98/254 - Day 91 (N=38,106,144,84) | 8.46 [4.85 to 15] | 18 [13 to 24] | 14 [11 to 19] | 14 [10 to 18]

5. Primary Outcome: Percentages of Subjects With Four-fold Increases in hSBA Titers Against the Serogroup B Indicator Strains (H44/76, 5/99, and NZ98/254) and M10713 Strain.
Description: Antibody responses were assessed in terms of percentage of subjects achieving 4-fold increase in ELISA concentrations against vaccine antigen 287-953 on Day 91 over baseline (Day 1), following 2 doses of rMenB+OMV NZ, administered on Day 1 and Day 61.
Time Frame: Day 91 (one month after the second dose of the study vaccine).
Population: Analysis was done on Full Analysis Set
Measure: Number (95% Confidence Interval); unit: Percentage of Subjects
Arm/Group | CompDef | Asplenia | CompDef + Asplenia | Healthy
Number analyzed (Participants) | 39 | 105 | 144 | 85
Percentage of Subjects
  5/99 - Day 91 (N=37,103,140,82) | 92 [78.1 to 98.3] | 100 [96.5 to 100] | 98 [93.9 to 99.56] | 98 [91.5 to 99.70]
  H44/76 - Day 91 (N=39,104,143,84) | 87 [72.6 to 95.7] | 94 [87.9 to 97.9] | 92 [86.7 to 96.1] | 98 [91.7 to 99.71]
  M10713 - Day 91 (N=36,102,138,82) | 25 [12.1 to 42.2] | 33 [24.3 to 43.4] | 31 [23.6 to 39.6] | 33 [22.9 to 44.2]
  NZ98/254 - Day 91 (N=36,105,141,83) | 61 [43.5 to 76.9] | 80 [71.1 to 87.2] | 75 [67.2 to 82.1] | 73 [62.7 to 82.6]

6. Primary Outcome: Geometric Mean Concentrations (GMCs) of Antibodies Against Vaccine Antigen 287-953 Following a 2-dose Vaccination Schedule.
Description: Immune responses were measured as Enzyme-linked Immunosorbent Assay (ELISA) GMCs of antibodies against vaccine antigen 287-953 following 2 doses of rMenB+OMV NZ, administered on Day 1 and Day 61.
Time Frame: Day 1 and Day 91 (one month after the second dose of the study vaccine).
Population: Analysis was done on Full Analysis Set
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | CompDef | Asplenia | CompDef + Asplenia | Healthy
Number analyzed (Participants) | 40 | 106 | 146 | 84
IU/mL
  287-953 - Day 1 (N=39,106,145,84) | 33 [25 to 43] | 25 [21 to 29] | 27 [23 to 31] | 27 [23 to 31]
  287-953 - Day 91 (N=40,106,146,84) | 2039 [1436 to 2894] | 3418 [2780 to 4202] | 2973 [2492 to 3546] | 2957 [2450 to 3570]

7. Primary Outcome: ELISA GMRs of Antibodies Against Vaccine Antigen 287-953 Following a 2-dose Vaccination Schedule.
Description: Immune responses were measured as ELISA GMRs of antibodies against vaccine antigen 287-953 following 2 doses of rMenB+OMV NZ, administered on Day 1 and Day 61.
Time Frame: Day 1 and Day 91 (one month after the second dose of the study vaccine).
Population: Analysis was done on Full Analysis Set
Measure: Geometric Mean (95% Confidence Interval); unit: Ratios
Arm/Group | CompDef | Asplenia | CompDef + Asplenia | Healthy
Number analyzed (Participants) | 39 | 106 | 145 | 84
Ratios | 62 [40 to 97] | 138 [107 to 178] | 112 [90 to 193] | 111 [88 to 140]

8. Primary Outcome: Percentage of Subjects With Four-fold Increases in ELISA Concentrations Against the Vaccine Antigen 287-953.
Description: as for outcome 5
Time Frame: Day 91 (one month after the second dose of the study vaccine).
Population: Analysis was done on Full Analysis Set
Measure: Number (95% Confidence Interval); unit: Percentage of Subjects
Arm/Group | CompDef | Asplenia | CompDef + Asplenia | Healthy
Number analyzed (Participants) | 39 | 106 | 145 | 84
Percentage of Subjects | 97 [86.5 to 99.4] | 98 [93.4 to 99.77] | 98 [94.1 to 99.57] | 98 [91.7 to 99.71]

9. Secondary Outcome: Number of Subjects Reporting Solicited Local and Systemic AEs.
Description: Reactogenicity was presented in terms of percentages of subjects reporting solicited local and systemic AEs and other indicators.
Time Frame: From Day 1 until Day 7 after any vaccination.
Population: Analysis was done on Solicited Safety Set (all subjects in the exposed set with any solicited AE data).
Measure: Number; unit: participants
Groups:
- Total: Total of subjects
Arm/Group | CompDef | Asplenia | CompDef + Asplenia | Healthy | Total
Number analyzed (Participants) | 28 | 100 | 128 | 74 | 202
participants
  Any (< 6 years; N=12,9,21,13,34) | 12 | 8 | 20 | 13 | 33
  Any Local (< 6 years; N=12,9,21,13,34) | 12 | 6 | 18 | 12 | 30
  Any Systemic (< 6 years; N=12,9,21,13,34) | 11 | 6 | 17 | 12 | 29
  Any (≥ 6 years) | 27 | 98 | 125 | 74 | 199
  Any Local (≥ 6 years) | 26 | 98 | 124 | 74 | 198
  Any Systemic (≥ 6 years) | 21 | 75 | 96 | 60 | 156
  Erythema (< 6 years; N=12,9,21,13,34) | 7 | 4 | 11 | 6 | 17
  Induration (< 6 years; N=12,9,21,13,34) | 5 | 4 | 9 | 5 | 14
  Swelling (< 6 years; N=12,9,21,13,34) | 6 | 4 | 10 | 6 | 16
  Tenderness (<6 years; N=12,9,21,13,34) | 12 | 6 | 18 | 12 | 30
  Change in Eating Habits (<6 years;N=12,9,21,13,34) | 5 | 1 | 6 | 8 | 14
  Diarrhea (< 6 years; N=12,9,21,13,34) | 5 | 3 | 8 | 3 | 11
  Irritability (< 6 years; N=12,9,21,13,34) | 6 | 2 | 8 | 9 | 17
  Persistent Crying (< 6 years; N=12,9,21,13,34) | 2 | 2 | 4 | 6 | 10
  Rash (< 6 years; N=12,9,21,13,34) | 3 | 0 | 3 | 0 | 3
  Sleepiness (< 6 years; N=12,9,21,13,34) | 7 | 3 | 10 | 5 | 15
  Vomiting (< 6 years; N=12,9,21,13,34) | 2 | 0 | 2 | 0 | 2
  Fever (≥38°C) (< 6 years; N=12,9,21,13,34) | 3 | 1 | 4 | 4 | 8
  Prevention Pain/Fever (<6 years; N=12,9,21,13,34) | 5 | 1 | 6 | 4 | 10
  Treat. P/F (< 6 years; N=12,9,21,13,34) | 5 | 3 | 8 | 11 | 19
  Erythema (≥ 6 years) | 7 | 19 | 26 | 27 | 53
  Induration (≥ 6 years) | 11 | 27 | 38 | 19 | 57
  Swelling (≥ 6 years) | 8 | 24 | 32 | 24 | 56
  Pain (≥ 6 years) | 25 | 97 | 122 | 71 | 193
  Arthralgia (≥ 6 years) | 7 | 25 | 32 | 18 | 50
  Fatigue (≥ 6 years) | 11 | 55 | 66 | 46 | 112
  Headache (≥ 6 years) | 11 | 47 | 58 | 35 | 93
  Myalgia (≥ 6 years; N=28,100,128,73,201) | 8 | 31 | 39 | 27 | 66
  Nausea (≥ 6 years) | 7 | 28 | 35 | 15 | 50
  Rash (≥ 6 years) | 7 | 9 | 16 | 6 | 22
  Fever (≥ 38°C) (≥ 6 years) | 6 | 6 | 12 | 5 | 17
  Prev. Pain/Fever (≥ 6 years) | 5 | 9 | 14 | 15 | 29
  Treat. Pain/Fever (≥ 6 years) | 14 | 39 | 53 | 38 | 91

10. Primary Outcome: Number Of Subjects With Unsolicited Adverse Events (AEs).
Description: Safety was assessed as the number of subjects who reported unsolicited AEs collected from Day1 through Day 7 after any vaccination; serious adverse events (SAEs), AEs leading to withdrawal and medically attended AEs were collected throughout the study period (Day1-Day 91).
Time Frame: At Day1 through Day 7 after any vaccination and throughout the study period (Day 1 to Day 91)
Population: Analysis was done on the Unsolicited Safety Set (all subjects in the exposed set with postvaccination unsolicited AE records).
Measure: Number; unit: participants
Arm/Group | CompDef | Asplenia | CompDef + Asplenia | Healthy
Number analyzed (Participants) | 40 | 110 | 150 | 87
participants
  Any AE | 17 | 38 | 55 | 34
  At least possibly related AEs | 9 | 19 | 28 | 18
  Any SAEs | 1 | 5 | 6 | 0
  At least Possibly Related SAEs | 0 | 0 | 0 | 0
  AEs Leading to Death | 0 | 0 | 0 | 0
  AEs Leading to Withdrawal | 0 | 1 | 1 | 0
  Medically Attended AEs | 13 | 26 | 39 | 18

ADVERSE EVENTS:
Time Frame: Throughout the entire study period (Day 1 to Day 91)
Groups:
- CompDef: Subjects aged ≥ 2 to ≤17 years with complement deficiencies received 2 doses of rMenB+OMV NZ administered 2 months apart.
- CompDef + Asplenia: Subjects aged ≥ 2 to ≤17 years with either complement deficiencies or Asplenia received 2 doses of rMenB+OMV NZ administered 2 months apart.
- Total: Total number of Subjects
Arm/Group | CompDef | Asplenia | CompDef + Asplenia | Healthy | Total
Serious Adverse Events (participants affected / at risk) | 1/40 | 5/110 | 6/150 | 0/87 | 6/237
Other Adverse Events (participants affected / at risk) | 39/40 | 106/110 | 145/150 | 87/87 | 232/237
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CompDef (N=40) | Asplenia (N=110) | CompDef + Asplenia (N=150) | Healthy (N=87) | Total (N=237)
INTRACARDIAC THROMBUS (Cardiac disorders) | 0 | 1 | 1 | 0 | 1
APPENDICITIS (Infections and infestations) | 0 | 1 | 1 | 0 | 1
GASTROENTERITIS SALMONELLA (Infections and infestations) | 0 | 1 | 1 | 0 | 1
RESPIRATORY TRACT INFECTION VIRAL (Infections and infestations) | 1 | 0 | 1 | 0 | 1
TONSILLITIS (Infections and infestations) | 0 | 1 | 1 | 0 | 1
CONCUSSION (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 1
RESPIRATORY DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CompDef (N=40) | Asplenia (N=110) | CompDef + Asplenia (N=150) | Healthy (N=87) | Total (N=237)
DIARRHOEA (Gastrointestinal disorders) | 5 | 4 | 9 | 4 | 13
NAUSEA (Gastrointestinal disorders) | 7 | 28 | 35 | 15 | 50
VOMITING (Gastrointestinal disorders) | 3 | 0 | 3 | 0 | 3
CRYING (General disorders) | 2 | 2 | 4 | 6 | 10
FATIGUE (General disorders) | 11 | 55 | 66 | 46 | 112
INJECTION SITE ERYTHEMA (General disorders) | 15 | 23 | 38 | 34 | 72
INJECTION SITE INDURATION (General disorders) | 17 | 32 | 49 | 26 | 75
INJECTION SITE PAIN (General disorders) | 37 | 103 | 140 | 83 | 223
INJECTION SITE SWELLING (General disorders) | 14 | 28 | 42 | 32 | 74
PYREXIA (General disorders) | 10 | 7 | 17 | 10 | 27
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 7 | 25 | 32 | 18 | 50
MYALGIA (Musculoskeletal and connective tissue disorders) | 8 | 31 | 39 | 27 | 66
HEADACHE (Nervous system disorders) | 11 | 48 | 59 | 35 | 94
SOMNOLENCE (Nervous system disorders) | 7 | 3 | 10 | 5 | 15
EATING DISORDER (Psychiatric disorders) | 5 | 1 | 6 | 8 | 14
IRRITABILITY (Psychiatric disorders) | 7 | 2 | 9 | 9 | 18
RASH (Skin and subcutaneous tissue disorders) | 10 | 9 | 19 | 6 | 25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreement with its investigators may vary.

However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publications of the pooled data (i.e., data from all sites) in the clinical trial.